CLINICAL TRIAL: NCT05772429
Title: Long-term Follow-up of a Multicentre, Non-interventional, Prospective Cohort of Participants Prescribed Epidyolex in France in a Real-life Setting
Brief Title: Long-Term Follow-Up of a Cohort of Participants Prescribed Epidyolex in France in a Real-life Setting
Acronym: OPERA
Status: Active, not recruiting | Type: Observational
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: GWEP20125
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Seizures
Keywords: Seizure Therapy; Cannabidiol; GW CBD; Epidyolex; Epidiolex; Jazz CBD
MeSH Terms: conditions — Seizures | interventions — Cannabidiol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Epidyolex: Participants will receive Epidyolex in accordance with their routine clinical practice as prescribed by their physician.
  Interventions: Drug: Epidiolex

INTERVENTIONS:
Drug: Epidiolex — Administered as an oral solution
  Other Names: Cannabidiol; Epidyolex

SUMMARY:
This is a multi-center, non-interventional and prospective study of patients receiving Epidyolex as part of standard clinical practice in France. The study will state an overview of patient characteristics and clinical history (including age, sex, diagnosis, duration of epilepsy, predominant seizure type, previous medications, current co-medications and Epidyolex dose), and an evaluation of retention rates, safety profile, seizure activity, changes in executive function and quality of life measured in a 2-year follow-up period.

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals for whom treatment with Epidyolex has been initiated by a physician with experience in the treatment of epilepsy.
* The participant and/or parent(s)/legal representative is willing and able to give informed consent/assent for participation in the study.

Key Exclusion Criteria:

* Previously initiated with Epidyolex before the start of the study (especially during the French early access program (EAP)).

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants for whom Epidyolex is prescribed according to the approved therapeutic indications and criteria of the summary of product Characteristics (SmPC). Participants will be recruited from approximately 15 facilities specializing in treating rare epilepsies in France.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Retention Rate Percentage After Initiation of Treatment With Epidyolex | Up to 24 months post-dose.
  Retention rate will be measured through assessing the frequency of seizures and the length of time on treatment before a seizure event.

SECONDARY OUTCOMES:
Percent Change From Baseline in Seizure Frequency (Average Per 28 Days) | Up to 24 months post-dose.
50% Responder Rate | Up to 24 months post-dose.
75% Responder Rate | Up to 24 months post-dose.
100% Responder (Seizure Freedom) Rate | Up to 24 months post-dose.
Number of Seizure-Free Days (Average Per 28 Days) | Up to 24 months post-dose.
Longest Duration of Seizure-Free Days in the Last 28 Days | Up to 24 months post-dose.
Change From Baseline in Behavior Rating Inventory of Executive Function, Preschool Version (BRIEF-P) Score in Participants Aged ≤5 Years | Baseline; Up to 24 months post-dose.
  The BRIEF-P is a 63-item questionnaire which consists of a single Rating Form used by parents, teachers, and day care providers to assess a child's executive functions within the context of their everyday environments--home and preschool. High scores obtained on the BRIEF-P suggest a higher level of dysfunction in a specific domain of executive functions. The BRIEF rating scores is an ordinal set of a technically summarized degree of disorder in functionality: Never = 1 (Minimum), Sometimes = 2 and Often = 3 (Maximum).
Change From Baseline in Behavior Rating Inventory of Executive Function (BRIEF) Score in Participants Aged 6 to 18 Years | Baseline; Up to 24 months post-dose.
  BRIEF is an 86-item questionnaire used to assess the executive function behaviors at home and at school for children and adolescents ages 5-18. High scores obtained on the BRIEF suggest a higher level of dysfunction in a specific domain of executive functions. The BRIEF rating scores is an ordinal set of a technically summarized degree of disorder in functionality: Never = 1 (Minimum), Sometimes = 2 and Often = 3 (Maximum).
Change From Baseline in Behavior Rating Inventory of Executive Function, Adult Version (BRIEF- A) Score in Participants Aged >18 Years | Baseline; Up to 24 months post-dose.
  BRIEF-A is a patient-reported scale to measure various aspects of adult executive functioning and self-regulation in the person's everyday environment. It is a 75-item questionnaire that participants rate on a 3-point Likert scale (1 = behavior is never observed to 3 = behavior is often observed). Higher scores indicate greater impairment in executive functioning.
Modal Dose of Epidyolex Administered to Participants | Up to 24 months post-dose.
Maximum Dose of Epidyolex Administered to Participants | Up to 24 months post-dose.
Change from Baseline in Average Daily Dosage of Concomitant Anti-Epileptic Drugs (AEDs) and Other Medicines | Up to 24 months post-dose.
Use of Rescue Medication Per Month | Up to 24 months post-dose.
  A month is defined as 28 days.
Physician Global Clinical Impression of Change (PGIC) Score | Up to 24 months post-dose.
  The PGIC comprises the following question: "Please assess the change in the patient's general functional abilities since enrollment," scored on a seven-point scale from 1 (Very Much Improved) to 7 (Very Much Worse). Lower scores on the scale indicate a better quality of life.
Caregiver Global Impression of Change (CGIC) Score | Up to 24 months post-dose.
  The CGIC comprises of the following question: "Since your child started treatment, please assess the status of your child's overall condition (comparing their condition now to their condition before treatment)," scored on a seven-point scale from 1 (Very Much Improved) to 7 (Very Much Worse). Lower scores on the scale indicate a better quality of life.
Change from Baseline in Health Utility Index Mark II (HUI-2) Score | Up to 24 months post-dose.
  The HUI-2 is a generic measure of health status and health-related quality of life. There are 15 questions in the questionnaire with 1-week recall completed by the caregiver. Answers to the questionnaire are mapped into a classification system of 7 sets of utility scores (sensation, mobility, emotion, cognition, self-care, pain, and fertility) with a scoring scale of a minimum score of 0.00 (lack of functional capacity or most disabled) to a maximum of 1.00 (full function or no disability). A higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Locations (29):
- France (29):
  - CHU Amiens-service adulte, Amiens
  - CHU Amiens-service enfant, Amiens
  - CHU Angers - service adulte, Angers
  - CHU Angers - service enfant, Angers
  - CHU Bordeaux - service adulte, Bordeaux
  - CHU Bordeaux,neuropédiatrie, Bordeaux
  - GH Est - Hôpital Femme Mère Enfant, Bron
  - HCL - Lyon - service adulte, Bron
  - CHU Dijon - service neurophysiologie clinique, Dijon
  - CHU Grenoble - service adulte, Grenoble
  - CHU Grenoble - service enfant, Grenoble
  - APHP Kremlin Bicetre - service enfant, Le Kremlin-Bicêtre
  - CHU Lille - service enfant, Lille
  - Hôpital Salengro - service adulte, Lille
  - APHM - Marseille - service adulte, Marseille
  - Hôpital de la Timone - service enfant, Marseille
  - CHU Nancy - service adulte, Nancy
  - CHU Nancy - service enfant, Nancy
  - APHP Pitié Salpetriere- service adulte, Paris
  - APHP Robert Debré - service enfant, Paris
  - APHP Necker - service enfant, Paris
  - CHU Rennes - service adulte, Rennes
  - CHU Rennes - service enfant, Rennes
  - CHU Strasbourg - service enfant, Strasbourg
  - Hôpital de Hautepierre - service adulte, Strasbourg
  - CHU Toulouse - service adulte, Toulouse
  - CHU Toulouse - service enfant, Toulouse
  - Hôpital Bretonneau - service adulte, Tours
  - Hôpital Clocheville - service enfant, Tours